CLINICAL TRIAL: NCT03771677
Title: A Clinical Controlled Study to Optimize the Therapeutic Pathway of Peginterferon Alfa-2b Treatment in Patients With Chronic Hepatitis B Based on IFNA2p.Ala120Thr /ISGs Gene Spectrum.
Brief Title: To Optimize the Therapeutic Pathway of Peginterferon Treatment in Patients With CHB Based on IFNA2p.Ala120Thr /ISGs.
Acronym: IFNA2/ISGs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First People's Hospital of Foshan (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chan Xie, Professor of department of infectious disease Third Affiliated Hospital,Sun Yat-Sen University, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XC1
Record Dates: First submitted 2018-12-08; First posted 2018-12-11 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Hepatitis B
Keywords: Chronic Hepatitis B; IFNA2p.Ala120Thr /ISGs
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — Nucleotides; Interferon alpha-2; peginterferon alfa-2a

STUDY DESIGN:
Intervention Model Description: Drug: nucleotide analogues(NAs)
  Drug: Peginterferon alfa-2a and nucleotide analogues(NAs)
Masking Description: Active Comparator:nucleotide analogues(NAs) patients continue to use NAs
  Experimental: peg-interferon alfa-2a patients switch to sequential peg-interferon α-2a
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator:NAs group (Active Comparator): Active Comparator:nucleotide analogues(NAs)
  patients continue to use NAs
  Interventions: Drug: Nucleotide Analog
- Experimental:PEG-IFN group (Experimental): Experimental: peg-interferon alfa-2a
  patients use peg-interferon α-2a and nucleotide analogues(NAs)
  Interventions: Drug: Nucleotide Analog; Drug: Interferon Alfa-2A

INTERVENTIONS:
Drug: Nucleotide Analog — such as Entecavir,entecavir 0.5mg per day
  Other Names: Nucleotide Analogs
Drug: Interferon Alfa-2A — Peginterferon alfa-2a 180ug per week
  Other Names: Pegasys
  Arms: Experimental:PEG-IFN group

SUMMARY:
The study is to guide clinical cure of peginterferon alfa-2a treatment in patients with chronic hepatitis B based on the detection of interferon gene mutation (IFNA2p.Ala120Thr) and interferon-stimulated genes (ISGs) detection gene spectrum.

DETAILED DESCRIPTION:
It is estimated that more than 400 million people are infected with hepatitis B virus (HBV) globally.How to make more patients with chronic hepatitis B get clinical treatment through the existing anti-viral treatment is an urgent problem to be solved.This study is a random, multi-center and open experiment,the collaborators includes the second people's hospital of zhongshan city, the eighth people's hospital of guangzhou city, and the first people's hospital of foshan city.

Patients with chronic hepatitis B who were treated with NAs for over 1 year,HBsAg quantification≤1500 IU/mL, HBeAg negative and serum HBV DNA quantification <100 IU/mL were enrolled in this study. In our study, the enrolled patient's IFNA2p.Ala120Thr without variation and ISGs>0.05 were divided into two groups. After informed consent , patients were grouped according to their treatment intentions,in one group, patients continued NAs for another 48 weeks. In another group , patients were treated with peg-interferon-2a and NAs for 48 weeks.Patient's BMI, genotype, family history, smoking history, drinking history, other medical history, suspected transmission channels, types and time of use were recorded in this study.Moreover, Patients were assessed every 12 weeks,included liver and kidney function, blood routine, HBV cccDNA, HBeAg quantification, HBsAg quantification, pgRNA and so on.In addition,liver imaging examination and liver hardness test were assessed every six months.

In this study, we will analyze whether clinical cure rates differed between patients with chronic hepatitis B treated with peginterferon alfa-2a and NAs;Bisedes,the baseline interferon variant site variants and changes in interferon-stimulated gene profile expression were analyzed to determine whether they could be used as molecular markers to predict clinical cure with interferon.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years old;
* HBsAg positive, HBsAg quantification≤1500 IU/mL;
* Serum HBV DNA quantification <100 IU/mL;
* HBeAg negative.

Exclusion Criteria:

* Treated with interferon in the past six months;
* Liver cirrhosis or HCC and other associated tumors;
* Women during pregnancy or lactation;
* With liver disease caused by other causes;
* Combination infection of HIV or other immunodeficiency diseases;
* With diabetes, autoimmune diseases and other organ dysfunction or failure;
* Combination of other serious complications (infection, hepatic encephalopathy,gastrointestinal bleeding, hepatorenal syndrome, etc.);
* Others who cannot be treated with interferon;
* Anyone cannot return to the hospital for follow-up and follow-up visits regularly as planned

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
HBsAg clearance rate | 48 weeks
  Whether the HBsAg clearance rate of patients who received interferon treatment was higher than those treated with nucleoside drugs.

SECONDARY OUTCOMES:
HBV cccDNA and pgRNA quantification dynamic change | 48 weeks
  The difference in cccDNA and pgRNA clearance rate between the two groups after 48 weeks of treatment in immune-controlled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Chan Xie, Principal Investigator — The Third Affliated Hospital of Sun Yat-sen University
Locations (1):
- Chan Xie, Guangzhou, Guangdong, China